CLINICAL TRIAL: NCT01120041
Title: Community-based Intergenerational Oral Health Promotion In Rural America
Brief Title: Community-based Intergenerational Oral Health Study
Acronym: Baby Smiles
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Christine Riedy and Philip Weinstein, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 37124-C; 5U54DE019346 (NIH); 09-016E
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Preventive Health Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prenatal MI - Postpartum MI (Experimental): Motivational interviewing counseling given during the prenatal and postpartum phases
  Interventions: Behavioral: motivational interviewing counseling
- Prenatal MI - Postpartum Health Ed (Experimental): Motivational interviewing counseling given during the prenatal phase with traditional health education given during the postpartum phase
  Interventions: Behavioral: motivational interviewing counseling
- Prenatal Health Ed - Postpartum MI (Experimental): Traditional health education given during the prenatal phase with motivational interviewing counseling given during the postpartum phase
  Interventions: Behavioral: motivational interviewing counseling
- Prenatal Health Ed/Postpartum Health Ed (Placebo Comparator): Traditional health education given during the prenatal phase and the postpartum phase
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: motivational interviewing counseling — Motivational interviewing counseling given during the prenatal and postpartum phases
  Arms: Prenatal MI - Postpartum MI
Behavioral: motivational interviewing counseling — Motivational interviewing counseling given during the prenatal phase with traditional health education given during the postpartum phase
  Arms: Prenatal MI - Postpartum Health Ed
Behavioral: motivational interviewing counseling — Traditional health education given during the prenatal phase with motivational interviewing counseling given during the postpartum phase
  Arms: Prenatal Health Ed - Postpartum MI
Behavioral: health education — Traditional health education given during the prenatal phase and the postpartum phase
  Arms: Prenatal Health Ed/Postpartum Health Ed

SUMMARY:
The purpose of this study is to determine whether giving brief motivational interviewing counseling during the prenatal and/or postnatal period(s) will increase utilization of preventive dental care and improve the oral health of rural, low-income pregnant and postpartum women and their children, and to increase the number of home oral health practices taken by these women to prevent caries in their young children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (week 26 or earlier)
* At least 15 years of age
* Medicaid eligible
* Speaks English
* Willing and able to comply with study instructions
* Mother AND child available for length of the study (~ 24 months)

Exclusion Criteria:

-

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Visiting the dentist during pregnancy and up to two months postpartum for the mother and visiting the dentist before 18 months for the child. | During pregnancy and up to two months post partum (mother); up to 18 months (child)

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Riedy, PhD, MPH, Principal Investigator — University of Washington; Philip Weinstein, PhD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - Josephine County Public Health Department, Grants Pass, Oregon
  - Jefferson County Public Health Department, Madras, Oregon
  - Lincoln County Human Services Department, Newport, Oregon
  - Douglas County Health & Social Services, Roseburg, Oregon

REFERENCES:
- [Derived] Riedy CA, Weinstein P, Mancl L, Garson G, Huebner CE, Milgrom P, Grembowski D, Shepherd-Banigan M, Smolen D, Sutherland M. Dental attendance among low-income women and their children following a brief motivational counseling intervention: A community randomized trial. Soc Sci Med. 2015 Nov;144:9-18. doi: 10.1016/j.socscimed.2015.09.005. Epub 2015 Sep 8. PMID 26372934
- [Derived] Weinstein P, Milgrom P, Riedy CA, Mancl LA, Garson G, Huebner CE, Smolen D, Sutherland M, Nykamp A. Treatment fidelity of brief motivational interviewing and health education in a randomized clinical trial to promote dental attendance of low-income mothers and children: Community-Based Intergenerational Oral Health Study "Baby Smiles". BMC Oral Health. 2014 Feb 24;14:15. doi: 10.1186/1472-6831-14-15. PMID 24559035
- [Derived] Milgrom P, Riedy CA, Weinstein P, Mancl LA, Garson G, Huebner CE, Smolen D, Sutherland M. Design of a community-based intergenerational oral health study: "Baby Smiles". BMC Oral Health. 2013 Aug 6;13:38. doi: 10.1186/1472-6831-13-38. PMID 23914908